CLINICAL TRIAL: NCT02547142
Title: Evaluation of the Implementation of an Early Integrated Palliative Care Program in the Esophageal Cancer Population
Brief Title: Early Integration of Palliative Care in Esophageal Cancer Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study futility with regards to recruitment
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SJHH_EarlyPalliativeCare_EDAP
Record Dates: First submitted 2015-08-28; First posted 2015-09-11 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Esophageal Cancer
Keywords: Prospective Pre-Post Evaluation; Early Palliative care; FACT-E questionnaire; HADS questionnaire; Patient Health Questionnaire-9 (PHQ-9)
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early Palliative Care Group (Experimental): This is the intervention group and will consist of patients that have been randomized into the early palliative group, with a consultation expected to take place within one week of randomization. Patients in this group will still receive appropriate guideline based oncologic care including any surgical, brachytherapy, chemotherapy or radiotherapy services, along with palliative services.
  Interventions: Other: Early Palliative Care

INTERVENTIONS:
Other: Early Palliative Care — Metastatic esophageal cancer patients that receive early palliative care along with standard oncological care

SUMMARY:
Palliative care physicians and nurses are trained to help reduce suffering and improve quality of life in patients under their care. Their services also include other components such as referral to dietitians, social workers and community resources, to assist patients in their homes. In addition to this, they may also administer interventions to make patients more comfortable, assisting them and their families in making important decisions and providing support, during that time.

At present, palliative care is provided to esophageal cancer patients on an as-needed basis, through the referral of a heath care professional or the patient's request. This study aims to assess the impact of the integration of early palliative care combined with appropriate medical care in the metastatic esophageal cancer population, so that patients can benefit from these services at an earlier stage. It is hoped that this will improve quality of life, symptom management, depression and anxiety, as well as survival.

DETAILED DESCRIPTION:
Previous reports suggest that starting palliative care early in patients with breast, colorectal, prostate and lung cancers appear to improve quality of life, symptom management, depression, anxiety and perhaps even survival, but it has never been tested in patients with esophageal cancer.This study aims to assess the impact of the introduction of early palliative care services on the esophageal cancer population, as opposed to traditional palliative care, which is provided on an as-needed basis, usually in end-of-life situations.

The study is a prospective one-armed pre-post intervention evaluation. Eligible patients that have consented will receive an early consultation with the palliative care group. In addition to this, the patients will be administered appropriate oncological care including surgical, brachytherapy, chemotherapy or radiotherapy services. The patients will be referred to the palliative service at the time of consent, with a consultation taking place within one week of referral receipt. The nurses and physicians involved in the palliative service will not only provide symptom management, psychosocial support, assistance with treatment related decisions and other patient needs. Information about symptoms, anxiety and depression, and quality of life will be collected through surveys at two timepoints - at baseline, when the patient consents and at 12 weeks post diagnosis of metastatic disease. The primary outcome of the study is the change in quality of life perceived by esophageal cancer patients at the two timepoints. Secondary outcomes include differences in esophageal cancer specific symptoms and anxiety and depression scores at the two timepoints, as well as patient survival information.

This study is integrated into the currently operational Esophageal Diagnostic Assessment Program (EDAP) conceptualized and implemented at St. Joseph's Healthcare Hamilton. It is hoped that this study will also help to establish the full integration of palliative care into the overall care of patients with esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly diagnosed or referred to the Esophageal Diagnostic Assessment Program (EDAP) program with suspicious findings found to be esophageal cancer AND
* Patients who present with metastatic disease, defined as N3 lymph node involvement or distant metastatic deposits as confirmed on PET scan
* Patients must have been notified by a member of their healthcare team of their prognosis and palliative categorization as noted in the patient chart within 8 weeks of diagnosis
* Patients may undergo esophagectomy, stenting, brachytherapy or palliative intent chemotherapy or radiotherapy as clinically indicated

Exclusion Criteria:

* Individuals unable to complete questionnaires with assistance
* Patients presently undergoing neoadjuvant chemotherapy or radiotherapy for malignancy
* Patients with recurrent esophageal cancer
* Patients who are referred back to EDAP for restaging after completing neoadjuvant therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-01-18 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Quality Of Life | As reported by questionnaire at 12 weeks after study consent
  Change in perceived quality of life as reported by esophageal cancer patients.

SECONDARY OUTCOMES:
Esophageal cancer-specific symptom score | As reported by questionnaire at 12 weeks after study consent
  Reported using the Functional Assessment of Cancer Therapy-Esophagus (FACT-E) tool - includes physical well-being, social/family well-being, emotional well-being, functional well-being, and symptom-specific measures. Scores range from 0 (not at all) to 4 (very much), and assesses how severely the symptom affects patients.
Esophageal cancer-specific symptom management score | As reported by questionnaire at 12 weeks after study consent
  The Patient Health Questionnaire (PHQ-9) will be used to measure the impact of the intervention on patient symptom management
Anxiety Score | As reported by questionnaire at 12 weeks after study consent
  Anxiety scores reported on the Hospital Anxiety and Depression Scale (HADS) Scale. The scores are summed to obtain a "normal", "borderline abnormal" or "abnormal" score
Depression Score | As reported by questionnaire at 12 weeks after study consent
  Depression scores reported on the Hospital Anxiety and Depression Scale (HADS) Scale. The scores are summed to obtain a "normal", "borderline abnormal" or "abnormal" score
Total duration of time from date of metastatic diagnosis to date of death | Time difference between date of diagnosis to the confirmed date of death as noted in patient medical records, assessed up to 60 months after the date of metastatic diagnosis
  Patient survival post metastatic esophageal cancer diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Christian Finley, MD MPH FRCSC, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No